CLINICAL TRIAL: NCT02746497
Title: The Efficacy of ACupuncture On Menopausal Symptoms (ACOM): A Randomized Controlled Trial
Brief Title: The Efficacy of ACupuncture On Menopausal Symptoms (ACOM)
Acronym: ACOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Research Unit Of General Practice, Copenhagen (Other); Danish Society for Evidence Based Acupuncture (DSEA) (Unknown); Idella Foundation (Unknown); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kamma Sundgaard Lund, Medical Doctor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1072031001
Record Dates: First submitted 2016-04-04; First posted 2016-04-21 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Menopause
Keywords: Menopause; Hot flushes; Acupuncture; Randomized controlled trial
MeSH Terms: conditions — Hot Flashes | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group E (early intervention) (Active Comparator): One weekly treatment with acupuncture in five consecutive weeks. In trial week 1-5 Group E will receive treatment and Group L will act as control group.
  Interventions: Procedure: Acupuncture
- Group L (late intervention) (Active Comparator): After trial week five the Groups must cross-over. Group L will then receive treatment for five weeks (trial week 6-11) and Group E will act as follow up group.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture style; Western Medical Acupuncture (WMA). In WMA all types of sham (placebo) acupuncture are believed to produce a certain amount of sensory stimulation and thereby a possible therapeutic effect. In addition, other studies have shown that sham acupuncture is associated with a moderately large nonspecific effect and compared to other inert placebo intervention the effect associated with sham acupuncture might be larger. Thus we use a control group instead of a placebo group.
  Needles; sterile disposable needles (Plandent) size 0.30x30mm. The needles will be inserted perpendicularly and rotated manual between finger and thumb for a few seconds to elicit "de-qi". Needle retention time will be 10 minutes. Afterward the needle will be removed. Acupuncture points; CV-3, CV-4, LR-8, SP-6, SP-9. In total 8 points as LR-8, SP-6, SP-9 are given bilaterally.

SUMMARY:
As a natural part of the menopause the ovaries production of sex hormones declines. This can lead to different menopausal related symptoms. About two-thirds of postmenopausal women experience hot flushes and 10-20% find these hot flushes very stressful.

The aim of this study is to determine and evaluate the efficacy of acupuncture on menopausal symptoms; in particular hot flushes. The study will be a randomized controlled trial. Primary outcome is change in hot flushes. Secondary outcome is change in other menopausal related symptoms.

DETAILED DESCRIPTION:
Hot flushes and night sweats are common menopausal symptoms. Around 75% of menopausal women experience hot flushes and 10-20% of all postmenopausal women find these hot flushes very stressful. Some menopausal women also experience other symptoms such as emotional vulnerability, sleeping problems, fatigue, joint pain, cognitive changes, vaginal dryness and loss of sexual desire.

On average women experience the menopause in the beginning of the early fifties. Menopausal symptoms are commonly experienced in 4-5 years and for some women even longer. Besides individual differences within a homogenous population the experience of menopausal symptoms also differs among different cultures and ethnic groups.

Hormone therapy (HT) has in many years been an effective treatment for menopausal symptoms. However, research has shown that long-term HT increases the risk of breast cancer and thromboembolic disorders. Other medications such as antidepressants or antiepileptics have been tried but are normally not recommended. Relaxation, exercise and use of different herbs have also been suggested but currently no convincing results. Hence, alternative effective treatments with few side effects are desired.

Acupuncture has in several studies shown an effect on menopausal hot flushes. However due to different study design, acupuncture style and outcome measures it is difficult to compare these studies. Moreover, many of these studies have been criticized for methodological errors and flaws e.g. poor design, lack of follow up, small sample size, inadequate control group, not standardized acupuncture points, problems with drop outs and blinding of the participants. Consequently, further research and more well-designed randomized controlled trials (RCTs) are needed.

It is estimated that approximately one-third of the general practitioners in Denmark on a regular basis are using acupuncture as part of their treatment of patients. A study from 2013 showed that about 20 % of the Danish hospital departments, distributed among 40% of the Danish hospitals, offered complementary and alternative medicine (CAM). Almost 70% of these treatments were acupuncture. Experience from this project could potentially kick start a research tradition of acupuncture, and lead to an expansion of an "evidence-based" use of acupuncture in the Danish health-care system.

HYPOTHESIS Treatment with acupuncture can reduce menopausal symptoms; in particular hot flushes.

AIM To determine and evaluate the efficacy of acupuncture on menopausal symptoms.

METHOD The study is designed as a randomized controlled trial and reporting will follow the STRICTA method which is an official extension of CONSORT statement.

RECRUITMENT AND SETTING Study subjects will primarily be recruited through general practitioners, the Danish Society for Evidence based Acupuncture (DSEA) and groups for menopausal women on social media.

The trial will take place in Danish primary care medical clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Woman
2. Age: 40-65 years
3. "Quite a bit" or "a lot" bothered by hot flushes (score ≥4 on a validated scale measuring hot flushes (MenoScores questionnaire (MSQ))
4. No conflicts of interests and have given oral and written consent
5. Must have an email address

Exclusion Criteria:

1. Hysterectomised and/or bilateral oophorectomised
2. Hormone therapy for menopausal symptoms within the past 4 weeks
3. Hormonal intrauterine device within the past 4 weeks
4. Treatment with antidepressants and/or antiepileptics within the past 4 weeks
5. Other medical treatment for hot flushes (e.g. clonidin) within the past 4 weeks
6. Other herbal remedies/alternative treatment for menopausal symptoms (e.g. Black Cohosh, Red Clover, Evening Primrose oil, Melbrosia) within the past 4 weeks
7. Alcohol consumption exceeding 21 drinks per week
8. Using prescribed sleeping pills and/or prescribed sedatives
9. Treatment with corticosteroids within the past 4 weeks (inhaled steroids not excluded)
10. Previously diagnosed with breast cancer, endometrial cancer, cervical cancer or ovarian cancer
11. Diagnosed with other severe cancer disease within the past 5 years
12. Heart valve disease
13. Insulin dependent and/or poorly controlled diabetes mellitus
14. Diagnosed with Thyroid disease
15. Under investigation for serious disease e.g. cancer
16. Pregnancy or breast-feeding within the past two years
17. Received acupuncture treatment within the past 6 months
18. Participating in another trial or participated in another trial in the past 2 weeks before screening

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Hot flushes (based on the hot flushes scale from MSQ) | 6 weeks
  Change in hot flushes from baseline to week 6 expressed by a score on the hot flushes scale from the MSQ.
  The MenoScores Questionnaire (MSQ) is developed and validated based on a literature review, 2 focus-groups, 4 single-interviews, 4 pilot-tests and a cross-sectional validation study where 1504 women answered a draft version of the questionnaire. Data collected in this validation study were analysed using Rasch models resulting in the MenoScores Questionnaire (MSQ), which encompasses 11 scales and 1 single item, measuring different dimension of menopausal symptoms.
  All study subjects (both Group E and L) will receive the MSQ by email in study week 0, 3, 6, 8, 11 and 26 and asked to answer within 1 or 2 days. The MSQ can be answered on computer or tablet. If responses are missing, reminders will be sent out. When receiving the planned acupuncture treatment the MSQ must be answered 1 or 2 days before the 3th treatment and 1 week after the 5th (the last) treatment.

SECONDARY OUTCOMES:
Change in other menopausal related symptoms, in particular day and night sweats and menopausal specific sleeping problems, also measured by scales from the MSQ. | 6 weeks
  The secondary outcomes and assessment of these will be as followed:
  Change in day-and-night-sweats assessed by a scale from the MSQ, Change in general sweating assessed by a scale from the MSQ, Change in menopausal specific sleeping problems assessed by a scale from the MSQ, Change in emotional symptoms assessed by a scale from the MSQ, Change in memory assessed by a scale from the MSQ, Change in skin-hair symptoms assessed by a scale from the MSQ, Change in physical symptoms assessed by a scale from the MSQ, Change in abdominal symptoms assessed by a scale from the MSQ, Change in urinary and vaginal symptoms assessed by a scale from the MSQ, Change in sexual symptoms assessed by a scale from the MSQ, Change in tiredness assessed by a single item from the MSQ.
  All measured as change from baseline at week 6.
Legacy effect. | 11 weeks
  Outcomes in week 11 express the legacy-effect of acupuncture treatment on menopausal related symptoms. Evaluated using the MSQ.
Long term outcome | 26 weeks
  Outcomes in week 26 express any possible longer-lasting effect. Evaluated using the MSQ.

CONTACTS AND LOCATIONS:
Overall Officials: Kamma S Lund, MD, Principal Investigator — Section of General Practice
Locations (1):
- Section of General Practice, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson HD. Menopause. Lancet. 2008 Mar 1;371(9614):760-70. doi: 10.1016/S0140-6736(08)60346-3. PMID 18313505
- [Background] Stearns V, Ullmer L, Lopez JF, Smith Y, Isaacs C, Hayes D. Hot flushes. Lancet. 2002 Dec 7;360(9348):1851-61. doi: 10.1016/s0140-6736(02)11774-0. PMID 12480376
- [Background] Avis NE, Crawford SL, Greendale G, Bromberger JT, Everson-Rose SA, Gold EB, Hess R, Joffe H, Kravitz HM, Tepper PG, Thurston RC; Study of Women's Health Across the Nation. Duration of menopausal vasomotor symptoms over the menopause transition. JAMA Intern Med. 2015 Apr;175(4):531-9. doi: 10.1001/jamainternmed.2014.8063. PMID 25686030
- [Background] Green R, Polotsky AJ, Wildman RP, McGinn AP, Lin J, Derby C, Johnston J, Ram KT, Crandall CJ, Thurston R, Gold E, Weiss G, Santoro N. Menopausal symptoms within a Hispanic cohort: SWAN, the Study of Women's Health Across the Nation. Climacteric. 2010 Aug;13(4):376-84. doi: 10.3109/13697130903528272. PMID 20136411
- [Background] Maclennan AH, Broadbent JL, Lester S, Moore V. Oral oestrogen and combined oestrogen/progestogen therapy versus placebo for hot flushes. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD002978. doi: 10.1002/14651858.CD002978.pub2. PMID 15495039
- [Background] Prentice RL, Manson JE, Langer RD, Anderson GL, Pettinger M, Jackson RD, Johnson KC, Kuller LH, Lane DS, Wactawski-Wende J, Brzyski R, Allison M, Ockene J, Sarto G, Rossouw JE. Benefits and risks of postmenopausal hormone therapy when it is initiated soon after menopause. Am J Epidemiol. 2009 Jul 1;170(1):12-23. doi: 10.1093/aje/kwp115. Epub 2009 May 25. PMID 19468079
- [Background] Pachman DR, Jones JM, Loprinzi CL. Management of menopause-associated vasomotor symptoms: Current treatment options, challenges and future directions. Int J Womens Health. 2010 Aug 9;2:123-35. doi: 10.2147/ijwh.s7721. PMID 21072305
- [Background] Daley A, MacArthur C, Mutrie N, Stokes-Lampard H. Exercise for vasomotor menopausal symptoms. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD006108. doi: 10.1002/14651858.CD006108.pub2. PMID 17943886
- [Background] Dodin S, Blanchet C, Marc I, Ernst E, Wu T, Vaillancourt C, Paquette J, Maunsell E. Acupuncture for menopausal hot flushes. Cochrane Database Syst Rev. 2013 Jul 30;2013(7):CD007410. doi: 10.1002/14651858.CD007410.pub2. PMID 23897589
- [Background] Borud EK, Alraek T, White A, Fonnebo V, Eggen AE, Hammar M, Astrand LL, Theodorsson E, Grimsgaard S. The Acupuncture on Hot Flushes Among Menopausal Women (ACUFLASH) study, a randomized controlled trial. Menopause. 2009 May-Jun;16(3):484-93. doi: 10.1097/gme.0b013e31818c02ad. PMID 19423996
- [Background] Zaborowska E, Brynhildsen J, Damberg S, Fredriksson M, Lindh-Astrand L, Nedstrand E, Wyon Y, Hammar M. Effects of acupuncture, applied relaxation, estrogens and placebo on hot flushes in postmenopausal women: an analysis of two prospective, parallel, randomized studies. Climacteric. 2007 Feb;10(1):38-45. doi: 10.1080/13697130601165059. PMID 17364603
- [Background] Venzke L, Calvert JF Jr, Gilbertson B. A randomized trial of acupuncture for vasomotor symptoms in post-menopausal women. Complement Ther Med. 2010 Apr;18(2):59-66. doi: 10.1016/j.ctim.2010.02.002. Epub 2010 Mar 23. PMID 20430288
- [Background] Smith CA, Carmady B. Acupuncture to treat common reproductive health complaints: An overview of the evidence. Auton Neurosci. 2010 Oct 28;157(1-2):52-6. doi: 10.1016/j.autneu.2010.03.013. Epub 2010 May 21. PMID 20483671
- [Background] MacPherson H, Altman DG, Hammerschlag R, Youping L, Taixiang W, White A, Moher D; STRICTA Revision Group. Revised STandards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA): Extending the CONSORT statement. J Evid Based Med. 2010 Aug;3(3):140-55. doi: 10.1111/j.1756-5391.2010.01086.x. PMID 21349059
- [Background] Linde K, Niemann K, Schneider A, Meissner K. How large are the nonspecific effects of acupuncture? A meta-analysis of randomized controlled trials. BMC Med. 2010 Nov 23;8:75. doi: 10.1186/1741-7015-8-75. PMID 21092261
- [Background] Prairie BA, Wisniewski SR, Luther J, Hess R, Thurston RC, Wisner KL, Bromberger JT. Symptoms of depressed mood, disturbed sleep, and sexual problems in midlife women: cross-sectional data from the Study of Women's Health Across the Nation. J Womens Health (Larchmt). 2015 Feb;24(2):119-26. doi: 10.1089/jwh.2014.4798. Epub 2015 Jan 26. PMID 25621768
- [Background] Bokmand S, Flyger H. Acupuncture relieves menopausal discomfort in breast cancer patients: a prospective, double blinded, randomized study. Breast. 2013 Jun;22(3):320-3. doi: 10.1016/j.breast.2012.07.015. Epub 2012 Aug 18. PMID 22906948
- [Background] Kim KH, Kang KW, Kim DI, Kim HJ, Yoon HM, Lee JM, Jeong JC, Lee MS, Jung HJ, Choi SM. Effects of acupuncture on hot flashes in perimenopausal and postmenopausal women--a multicenter randomized clinical trial. Menopause. 2010 Mar;17(2):269-80. doi: 10.1097/gme.0b013e3181bfac3b. PMID 19907348
- [Background] Skovgaard L, Cour SL, Kristensen M. Use of complementary and alternative medicine in Danish Hospitals as reported by charge nurses at department level. Journal of Hospital Administration wwwscieduca/jha; http://dxdoiorg/105430/jhav2n2p22. 2013;Vol 2, No 2.:22-6.
- [Background] Rosted P. Akupunktur: på naturvidenskabeligt grundlag: Klim; 2003.
- [Background] Mintziori G, Lambrinoudaki I, Goulis DG, Ceausu I, Depypere H, Erel CT, Perez-Lopez FR, Schenck-Gustafsson K, Simoncini T, Tremollieres F, Rees M. EMAS position statement: Non-hormonal management of menopausal vasomotor symptoms. Maturitas. 2015 Jul;81(3):410-3. doi: 10.1016/j.maturitas.2015.04.009. Epub 2015 Apr 22. PMID 25982505
- [Background] Rosted P. [The effect of acupuncture on musculoskeletal disorders]. Ugeskr Laeger. 2005 Sep 19;167(38):3573-7. Danish. PMID 16219184
- [Derived] Waldorff FB, Bang CW, Siersma V, Brodersen J, Lund KS. Factors associated with a clinically relevant reduction in menopausal symptoms of a standardized acupuncture approach for women with bothersome menopausal symptoms. BMC Complement Med Ther. 2021 Jan 13;21(1):29. doi: 10.1186/s12906-021-03208-2. PMID 33441145
- [Derived] Lund KS, Siersma V, Brodersen J, Waldorff FB. Efficacy of a standardised acupuncture approach for women with bothersome menopausal symptoms: a pragmatic randomised study in primary care (the ACOM study). BMJ Open. 2019 Feb 19;9(1):e023637. doi: 10.1136/bmjopen-2018-023637. PMID 30782712
- [Derived] Lund KS, Brodersen J, Siersma V, Waldorff FB. The efficacy of acupuncture on menopausal symptoms (ACOM study): protocol for a randomised study. Dan Med J. 2017 Mar;64(3):A5344. PMID 28260598